CLINICAL TRIAL: NCT07094139
Title: Clinical and Radiographic Outcomes of the JointMedica Custom-Made Resurfacing Device
Status: Not yet recruiting | Type: Observational
Sponsor: JointMedica Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CI003
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Real World Data; Safety and Effectiveness; Patient Reported Outcome (PRO)
Keywords: Custom-Made Hip Resurfacing; Hip Resurfacing; Hip Arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: The patient group is the entire group of patients who have been implanted with the JointMedica Custom-Made Hip Resurfacing system. This is the only group in the study, all patients will be assessed under the same criteria.

SUMMARY:
The Custom Resurfacing (CR) Implants are indicated for use for the reduction or relief of pain and/or improved hip function all skeletally mature patients where a total joint replacement is indicated, and where there is no other suitable, commercially distributed device available.

The Resurfacing System is a metal-on-polyethylene hip resurfacing device consisting of a metallic femoral component and an acetabular component made of Vitamin E HXLPE with a titanium coating on its bone-contacting surface.

The custom-Made Hip Resurfacing System is a single use device intended for hybrid fixation: cemented femoral head component and cementless acetabular component.

The goal of this observational study is to generate Real World Evidence (RWE) on the device performance of the Polymotion Hip Resurfacing (PHR) system and its use in patients who have been implanted with the device for the treatment of hip osteoarthritis.

This study will assess the following endpoints:

* The survivorship of the Acetabular Cup (Kaplan-Meier estimate) through 2 years of follow-up.
* Radiographic success of the implanted cups, through quantitative motion analysis to assess migration of the acetabular cups.
* Absence of subsequent surgical intervention at the acetabulum of there operated hip.
* Absence of serious, device-related adverse events.
* Patient reported outcomes through Harris Hip Score and SUSHI - UCLA Hip Score questionnaires.

DETAILED DESCRIPTION:
This is a retrospective and prospective study that will include a 41patients who were implanted with the JointMedica Custom-Made Hip Resurfacing device in the UK.

Patients will be invited to consent to participate in this study, which will require their attendance of a follow-up standard of care visit to gather clinical data on the safety and performance of their index hip, undergo an x-ray imaging and complete two questionnaires to assess their functionality and outcomes.

Patient data will be entered into electronic data capture systems and x-rays will be submitted to a core imaging laboratory, MMI, for analysis to assess the state and position of their acetabular cup.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above at the time of the surgery.
* Have had the JointMedica Custom-Made Hip Resurfacing device implanted between September 2020 to January 2025
* Written informed consent given by subject

Exclusion Criteria:

* There is no exclusion criteria for this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that underwent hip arthroplasty procedure with the JointMedica Custom-Made Hip Resurfacing device (V2.1+ Cup design) between September 2020 to January 2025.
  Subjects who have previously had the JointMedica Custom-Made Hip Resurfacing device implanted will be contacted to give consent to participate in the collection of additional follow-up visits described within this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acetabular Cup Survivorship | From the primary implantation to end through to 24 months and 27months+ post operation.
  The number of acetabular cups which are functional and not requiring additional surgical intervention following the primary implantation
Radiographic Success | Between primary implantation surgery and post-operative review at 24-months and 27+ months.
  Quantitative motion assessment of the acetabular cup at implantation and follow-up visit
Serious Device-Related Adverse Events | From primary implantation to post-operative visit at 24-months or 27+months
  Occurrence and severity of adverse events including necessitation of secondary surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Treacy, Principal Investigator
Locations (1):
- RBC Treacy Practice, Worcester, Bromsgrove, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes